CLINICAL TRIAL: NCT01628965
Title: An Open-label Long-term Extension Trial From Phase II/III of SPM962 (243-07-001) in Early Parkinson's Disease Patients With Non-concomitant Treatment of L-dopa
Brief Title: A Long-Term Extension Trial From Phase II/III of SPM 962 in Early Parkinson's Disease Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 243-07-002
Record Dates: First submitted 2012-06-25; First posted 2012-06-27 (Estimated); Results first posted 2014-03-19 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-02

CONDITIONS: Parkinson's Disease
Keywords: SPM 962; rotigotine; Parkinson's disease; monotherapy
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SPM 962 (Experimental): SPM 962 transdermal patch
  Interventions: Drug: SPM 962

INTERVENTIONS:
Drug: SPM 962 — SPM 962 transdermal patch once a daily up to 36.0 mg/day
  Other Names: rotigotine

SUMMARY:
Safety of SPM 962 in a once-daily repeated long-term treatment in Parkinson's disease patients who are not concomitantly treated with L-dopa will be investigated with a doses.

ELIGIBILITY:
Inclusion Criteria:

* Subject completed the preceding trial 243-07-001 (NCT00537485)

Exclusion Criteria:

* Subject discontinued from the preceding trial 243-07-001.
* Subject had a serious adverse event which association with the investigational drug was not ruled out during trial 243-07-001.
* Subject has a persistent serious adverse event at the baseline, which was observed and association with the investigational drug was ruled out during trial 243-07-001.
* Subject had persistent hallucination or delusion during trial 243-07-001.
* Subject has psychiatric conditions such as confusion, excitation, delirium, abnormal behaviour at the baseline.
* Subject has orthostatic hypotension or a systolic blood pressure (SBP) <= 100 mmHg and has a decrease of SBP from spine to standing position >= 30 mmHg at baseline.
* Subject has a history of epilepsy, convulsion etc. during trial 243-07-001.
* Subject develops serious ECG abnormality at the baseline.
* Subject has QTc-interval >= 500 msec at the baseline or subject has an increase of QTc-interval >= 60 msec from the baseline in the trial 243-07-001 and has a QTc-interval > 470 msec in female or > 450 msec in male at the baseline.
* Subject has a serum potassium level < 3.5 mEq/L at the end of the taper period in trial 243-07-001.
* Subject has a total bilirubin >= 3.0 mg/dL or AST(GOT) or ALT(GPT) greater than 2.5 times of the upper limit of the reference range (or >= 100 IU/L) at the end of the period in trial 243-07-001.
* Subject has BUN >= 30 mg/dL or serum creatinine >= 2.0 mg/dl at the end of the taper period in trial 243-07-001.
* Subject who plans pregnancy during the trial.
* Subject has dementia.
* Subject is unable to give consent.
* Subject is judged to be inappropriate for this trial by the investigator for the reasons other than above.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2008-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyoji Imaoka, Mr, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (7):
- Japan (7):
  - Chubu Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SPM 962
Started | 143
Completed | 94
Not Completed | 49
Not completed — Adverse Event | 30
Not completed — Lack of Efficacy | 7
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 1
Not completed — Discontinuation criteria | 8

BASELINE CHARACTERISTICS:
Arm/Group | SPM 962
Number analyzed (Participants) | 143
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 58
  >=65 years | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83
  Male | 60
Region of Enrollment [Number; unit: participants]
  Japan | 143

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Adverse Events, Vital Signs, and Laboratory Parameters
Description: Incidence and severity of adverse events, vital signs, and laboratory parameters up to 54 weeks after dosing.
  *decrease in difference between supine and standing systolic blood pressure
Time Frame: Up to 55 weeks after dosing
Population: Safety set (SS)
Measure: Number; unit: participants
Arm/Group | SPM 962
Number analyzed (Participants) | 143
participants
  Any AEs | 140
  Treatment-related AEs | 122
  SAEs | 18
  Severe AEs | 9
  Discontinuation due to AEs | 30
  Severe laboratory abnormality | 14
  ≥30 mmHg decrease* | 1
  Treatment-related AE of orthostatic hypotension | 2
  QTcB ≥500 ms | 1
  Weight decrease of 5% or more | 53
  Weight increase of 5% or more | 22

2. Secondary Outcome: Total of Unified Parkinson's Disease Rating Scale (UPDRS) Part 2 Sum Score and Part 3 Sum Score
Description: Mean change (LOCF) from baseline in Total of UPDRS Part 2 sum score and Part 3 sum up to 54 weeks after dosingUPDRS is a scale for monitoring Parkinson's Disease-related disability and impairment. The UPDRS consists of the following four sub-scales. Part 1: Mentation, Part 2: Activities of Daily Living, Part 3: Motor, Part 4: Complications. Part 2 assesses 13 items and Part 3 assesses 14 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: Baseline, Up to 54 weeks after dosing
Population: Full analysis set (FAS), last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM 962
Number analyzed (Participants) | 140
Scores on a scale
  Week 12 | -9.9 (8.7)
  Week 24 | -8.3 (9.5)
  Week 52 | -6.5 (10.1)

3. Primary Outcome: Skin Irritation Score of the Application Site
Description: Skin irritation score of the application site were evaluated according to the criteria below. The worst score throughout the treatment period was used in the analysis.
  -: no reaction, ±: mild erythema, +: erythema, ++: erythema and Oedema, +++: erythema and oedema and rash papular, or serous papule, or vesicles, ++++: bullosum
Time Frame: Up to 55 weeks after dosing
Population: SS
Measure: Number; unit: participants
Arm/Group | SPM 962
Number analyzed (Participants) | 142
participants
  - | 20
  ± | 57
  + | 46
  ++ | 12
  +++ | 6
  ++++ | 1
  +++> | 7

ADVERSE EVENTS:
Time Frame: 54 weeks
Arm/Group | SPM 962
Serious Adverse Events (participants affected / at risk) | 24/143
Other Adverse Events (participants affected / at risk) | 138/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPM 962 (N=143)
Positional Vertigo (Ear and labyrinth disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Gastric Ulcer Bleeding (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Gallbladder Polyp (Hepatobiliary disorders) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Altered State Of Consciousness (Nervous system disorders) | 1 (1)
Cerebral Infarction (Nervous system disorders) | 1 (1)
Disease Parkinson's (Nervous system disorders) | 1 (1)
Myoclonus (Nervous system disorders) | 1 (1)
Neuroleptic Malignant (Nervous system disorders) | 1 (1)
Delusion (Psychiatric disorders) | 1 (1)
Renal Impairment (Renal and urinary disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPM 962 (N=143)
Vertigo (Ear and labyrinth disorders) | 5 (6)
Nausea (Gastrointestinal disorders) | 47 (57)
Vomiting (Gastrointestinal disorders) | 22 (44)
Constipation (Gastrointestinal disorders) | 21 (21)
Application Site Reaction (General disorders) | 96 (100)
Oedema Peripheral (General disorders) | 7 (8)
Nasopharyngitis (Infections and infestations) | 26 (29)
Cystitis (Infections and infestations) | 5 (5)
Contusion (Injury, poisoning and procedural complications) | 7 (8)
Blood Creatine Phosphokinase Increased (Investigations) | 6 (7)
Back Pain (Musculoskeletal and connective tissue disorders) | 13 (13)
Dizziness (Nervous system disorders) | 8 (11)
Dyskinesia (Nervous system disorders) | 5 (7)
Somnolence (Psychiatric disorders) | 17 (18)
Insomnia (Psychiatric disorders) | 10 (10)
Hallucination (Psychiatric disorders) | 5 (7)
Hallucination Visual (Psychiatric disorders) | 5 (5)
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 5 (11)
Urticaria (Skin and subcutaneous tissue disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No